CLINICAL TRIAL: NCT02723110
Title: Defining the Physiological Mechanisms of Risk Genes for Hyperglycaemia, Insulin Resistance and Type 2 Diabetes
Acronym: DIVA - PAM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Oxford (Other)
Collaborators: University of Exeter (Other); Medical Research Council (Other Government)
Responsible Party: Sponsor
Other Study IDs: 15/SC/0072
Record Dates: First submitted 2016-02-12; First posted 2016-03-30 (Estimated); Last update posted 2016-06-22 (Estimated); Status verified 2016-06

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 Diabetes Risk
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Glucose Tolerance Test

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — EDTA plasma, serum, lithium heparin

GROUPS / COHORTS (2):
- rs78408340 heterozygous carriers
  Interventions: Other: 4 Hour Frequently Sampled Oral Glucose Tolerance Test; Other: Isoglycaemic Clamp
- homozygous non-risk allele carriers
  Interventions: Other: 4 Hour Frequently Sampled Oral Glucose Tolerance Test; Other: Isoglycaemic Clamp

INTERVENTIONS:
Other: 4 Hour Frequently Sampled Oral Glucose Tolerance Test — Blood glucose level(BGL) every 5 min, blood for hormone, biochemical analysis at -15,0,15,30,45,60,90,120,180, 240
  Other Names: OGTT
Other: Isoglycaemic Clamp — Glucose infusion over 4 hours to reproduce OGTT glucose curve to allow measurement of incretin effect. BGL every 5 min, blood for hormone, biochemical analysis at -15,0,15,30,45,60,90,120,180, 240
  Other Names: Matched clamp

SUMMARY:
Recent genetic association studies have identified variants in the Peptidyl-Glycine alpha-amidating mono-oxygenase (PAM) gene that increase the risk of diabetes likely through a defect in beta-cell function. This has been followed up and supported by novel kinetic assays and cellular studies. This investigation will recall heterozygous carriers of the risk allele at rs78408340 and age, BMI and gender matched controls from the Oxford Biobank. The study will compare the incretin effect, glucagon-like peptide-1(GLP-1), insulin, glucose levels and PAM protein activity in individuals both with and without the risk variant. The aim of the study is to gain mechanistic insight into the effect of the variant on human physiology and diabetes pathogenesis.

DETAILED DESCRIPTION:
Note: The study will utilize an adaptive study design with an interim analysis at 40 volunteers (20 v 20) with the possibility of adding an additional 20 volunteers to the study (10 v 10) if the criteria for futility or clear effect are not met.

The criteria are; stop and reject null hypothesis if t > 2.490 and stop and accept null hypothesis if t < 1.033. If the t falls between these values an additional 20 volunteers (10 v10) will be recruited. The decision to stop or additional volunteers will be based on the incretin effect (primary outcome).

ELIGIBILITY:
Inclusion Criteria:

* Adult, age 30-65 inclusive, healthy, appropriate genotype
* Mental capacity to consent

Exclusion Criteria:

* Demographics: <30 and >65 years old
* Medical history: Bariatric surgery, surgery on gut/ stomach; history of recent significant weight loss (>10% of weight in last year); known cardiovascular disease
* Medications: Currently prescribed glucose-lowering medication, oral/IV corticosteroid treatment, any medication effecting gastric motility or glucose metabolism

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers enrolled in the Oxford Biobank
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2015-06; Primary Completion 2016-07 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Calculated Incretin Effect | 3 months
  Will be calculated from the amount of IV glucose required to reproduce OGTT glycaemic profile

SECONDARY OUTCOMES:
Insulin concentration | 3 months
Glucose concentrations | 3 months
GLP-1 (glucagon-like peptide-1) amidated and unamidated concentration | 3 months
PAM enzyme activity assay | 3 months
  This assay is based off the protocol in the published literature, and is based on the turnover of radio-labelled substrate to quantify the amidating ability of the PAM enzyme

CONTACTS AND LOCATIONS:
Locations (1):
- OCDEM, University of Oxford, Oxford, Oxfordshire, United Kingdom